CLINICAL TRIAL: NCT03257891
Title: Multicenter, Prospective, Non-randomized, Phase II Trial Designed to Evaluate the Activity of Cabazitaxel in Patients With Advanced Adreno-Cortical- Carcinoma Progressing After Previous Chemotherapy Lines
Brief Title: Cabazitaxel Activity in Patients With Advanced AdrenoCortical-Carcinoma Progressing After Previous Chemotherapy Lines
Acronym: CabACC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP2729
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical Carcinoma; Cabazitaxel
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — cabazitaxel

STUDY DESIGN:
Intervention Model Description: A prospective, non-randomized, multicentre, open label, single arm, phase II study will be conducted in patients with advanced ACC treated with Cabazitaxel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): patients with advanced Adrenocortical- Carcinoma progressing after previous chemotherapy lines will be treated with Cabazitaxel
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel will be administered every 21 days

SUMMARY:
Adrenocortical cancer (ACC) is a rare aggressive tumor. The treatment of metastatic ACC is challenging and the current available treatments are mitotane, chemotherapy or the combination of both. Prognosis in locally advanced inoperable and metastatic ACC patients still remains poor, the 5-year overall survival being <15%. New treatment strategies are therefore needed. The taxanes are a class of drugs targeting the microtubules that have shown to be effective in the treatment of several malignancies but have not been fully developed in patients with ACC. Cabazitaxel is a new taxoid which promotes the tubulin assembly in vitro and stabilizes microtubules against cold-induced depolymerization as efficiently as docetaxel. Cabazitaxel was selected for development based on a better antiproliferative activity on resistant cell lines than docetaxel. The activity of the drug against several malignancies is currently tested in ongoing prospective studies, but to our knowledge neither preclinical nor clinical studies are currently testing cabaztaxel in ACC. This study is aimed to demonstrate that cabazitaxel is active in ACC, but the drug was never tested before in this clinical setting. A prospective, non-randomized, multicentre, open label, single arm, phase II study will be conducted in patients with advanced ACC. The phase II study will be conducted in 2 different Italian Institutions that are reference centers for ACC.

DETAILED DESCRIPTION:
CABAZITAXEL ADMINISTRATION Cabazitaxel will be administered at dose of 25 mg/m2 every 3 weeks, administered by IV route in 1 hour, for a maximum of 6 total cycles. The drug will be provided by Sanofi -Aventis S.p.A. Concomitant mitotane therapy will not be permitted however mitotane will be maintained in patients with hormone secreting tumors. Cycle length for cabazitaxel is 3 weeks. New cycles of therapy may not begin until Absolute Neutrophil Count (ANC) ≥1500/mm3, platelet count ≥75 000/mm3, and non-hematological toxicities (except alopecia) have recovered to baseline.

A maximum of 2 weeks delay is allowed between 2 treatment cycles.

PHARMACOKINETIC STUDY Another study aims will be to assess the toxicity of cabazitaxel therapy in ACC patients. As mitotane notoriously interfere with the metabolism of several drugs (11), an ancillary study will be conducted to assess the pharmacokinetic profile of cabazitaxel in the patient population with hormone secreting tumors that will maintain mitotane administration vs patients with non secreting ACC in which mitotane will be stopped. Blood samples will be collected in lithium heparinized tubes at fixed time points before and after drug infusion: Cycles 1 on Day 1 just before infusion, 30 min after start of infusion, 5 min before the end of 1-hour infusion (Tmax), 24 h, 48h and 96 h post-infusion. Cabazitaxel serum concentrations will be measured in plasma using a validated liquid chromatography-tandem mass spectrometry method: the Agilent 1260 Infinity LC equipped with an Agilent 6460 Triple Quadrupole Mass Spectrometer (QQQ) in electrospray mode systems.

STATISTICAL ANALYSIS All data collected at baseline, including recorded and derived variables will be described on all patients by means of summary descriptive statistics: mean, standard deviation, median, min, max, 25th and 75th percentiles for continuous variables; absolute and relative frequency for categorical variables. The relative frequencies will be calculated on the total patients with and without missing data. Whenever possible the data will be described by visit.

Chi square ore Fisher test, when applicable will be employed to compare categorical variables. Student T-test and analysis of variance for parametric or Wilcoxon's matched pairs signed-rank test and Friedman analysis of variance for non parametric data will be used to compare paired data. Simple correlation analysis will be performed by Spearman rho (coefficient of Spearman's rank correlation) for nonparametric distribution. Two-tailed tests will be used for all comparisons and p <0.05. All survival functions will computed using the Kaplan-Meier method. Survival curves will be compared with the log rank test.

CONCOMITANT MEDICATION Concurrent treatment with strong inhibitors and strong inducers of cytochrome P450 3A4 is not permitted. For patients who were receiving treatment with such agents, a 2-week washout period is required prior to randomization. Concurrent participation in another clinical trial or treatment with any other anti-cancer therapy is also not permitted. The Investigator may prescribe any other concomitant medications as deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC
* Locally advanced or metastatic disease not amenable to radical surgery resection
* Radiologically monitorised disease
* Progressing disease after one to three cytotoxic chemotherapy regimes (including a platin-based protocol)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy ≥ 3 months
* Age ≥ 18 years
* Adequate bone marrow reserve (neutrophils ≥ 1500/mm³ and platelets > 100.000/mm³)
* Effective contraception in pre-menopausal female and male patients
* Patient´s written informed consent
* Ability to comply with the protocol procedures
* Mitotane intake should be stopped one months before the study entry

Exclusion Criteria:

* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
* Serum creatinine > 1.5 x ULN or hepatic insufficiency, Hemoglobin <10.0 g/dL;
* Total bilirubin >1x ULN, Creatinine < 1.5 ULN;
* Decompensated heart failure (ejection fraction <45%), myocardial infarction or revascularization procedure during the last 6 months, unstable angina pectoris, uncontrolled cardiac arrhythmia
* Pregnancy or breast feeding
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Patients with serum levels of mitotane (evaluated one week before the study start) in the therapeutic range (14-20 mcg/ml).History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments) (see Annex 1 and Annex 2)
* Concomitant vaccination with yellow fever vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2021-01-24 (Estimated); Study Completion 2022-01-24 (Estimated)

PRIMARY OUTCOMES:
To assess the clinical benefit after 4 months of the cabazitaxel in patients with locally advanced or metastatic ACC who progressed after cytotoxic therapy. | 4 months
  CT scan evaluated according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Assessment of Objective Response Rates (ORR) | Every cycle (21 days) for a maximum of 6 cycles and for 6 months follow up. Total 1 year
  ORR evaluated by RECIST criteria
Assessment of overall survival | Every cycle (21 days) for a maximum of 6 cycles and for 6 months follow up. Total 1 year
  defined as the time from the date of the study start to date of death due to any cause
Assessment of quality of life | Every cycle (21 days) for a maximum of 6 cycles and for 6 months follow up. Total 1 year
  EORTC quality of life questionnaire (QLQ)-C30 will be administered to patients
Assessment of toxicity | Every cycle (21 days) for a maximum of 6 cycles and for 6 months follow up. Total 1 year
  evaluated by NCI CTCAE V4.03 criteria
Assessment of hormone response | Every cycle (21 days) for a maximum of 6 cycles and for 6 months follow up. Total 1 year
  Evaluation of adrenocorticotropic hormone (ACTH), Testosterone, Progesterone, Cortisol, (Deidroepiandrosterone) DHEA-S, 17-hydroxide- progesterone, Androstenedione in serum. Evaluation of 24 hours urinary cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, MD, Principal Investigator — Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Locations (1):
- Azienda Ospedaliera Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berruti A, Ferrero A, Sperone P, Daffara F, Reimondo G, Papotti M, Dogliotti L, Angeli A, Terzolo M. Emerging drugs for adrenocortical carcinoma. Expert Opin Emerg Drugs. 2008 Sep;13(3):497-509. doi: 10.1517/14728214.13.3.497. PMID 18764725
- [Result] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Result] Bates SE, Shieh CY, Mickley LA, Dichek HL, Gazdar A, Loriaux DL, Fojo AT. Mitotane enhances cytotoxicity of chemotherapy in cell lines expressing a multidrug resistance gene (mdr-1/P-glycoprotein) which is also expressed by adrenocortical carcinomas. J Clin Endocrinol Metab. 1991 Jul;73(1):18-29. doi: 10.1210/jcem-73-1-18. PMID 1675220
- [Result] Chen KG, Sikic BI. Molecular pathways: regulation and therapeutic implications of multidrug resistance. Clin Cancer Res. 2012 Apr 1;18(7):1863-9. doi: 10.1158/1078-0432.CCR-11-1590. Epub 2012 Feb 16. PMID 22344233
- [Result] Berruti A, Sperone P, Ferrero A, Germano A, Ardito A, Priola AM, De Francia S, Volante M, Daffara F, Generali D, Leboulleux S, Perotti P, Baudin E, Papotti M, Terzolo M. Phase II study of weekly paclitaxel and sorafenib as second/third-line therapy in patients with adrenocortical carcinoma. Eur J Endocrinol. 2012 Mar;166(3):451-8. doi: 10.1530/EJE-11-0918. Epub 2011 Dec 21. PMID 22189997
- [Result] Gradishar WJ, Tjulandin S, Davidson N, Shaw H, Desai N, Bhar P, Hawkins M, O'Shaughnessy J. Phase III trial of nanoparticle albumin-bound paclitaxel compared with polyethylated castor oil-based paclitaxel in women with breast cancer. J Clin Oncol. 2005 Nov 1;23(31):7794-803. doi: 10.1200/JCO.2005.04.937. Epub 2005 Sep 19. PMID 16172456
- [Result] Demeure MJ, Stephan E, Sinari S, Mount D, Gately S, Gonzales P, Hostetter G, Komorowski R, Kiefer J, Grant CS, Han H, Von Hoff DD, Bussey KJ. Preclinical investigation of nanoparticle albumin-bound paclitaxel as a potential treatment for adrenocortical cancer. Ann Surg. 2012 Jan;255(1):140-6. doi: 10.1097/SLA.0b013e3182402d21. PMID 22156929
- [Result] Mita AC, Figlin R, Mita MM. Cabazitaxel: more than a new taxane for metastatic castrate-resistant prostate cancer? Clin Cancer Res. 2012 Dec 15;18(24):6574-9. doi: 10.1158/1078-0432.CCR-12-1584. Epub 2012 Oct 22. PMID 23091116
- [Result] Montoya M, Brown JW, Fishman LM. Comparative effects of chemotherapeutic agents on the growth and survival of human adrenal carcinoma cells in culture. Horm Metab Res. 2008 May;40(5):302-5. doi: 10.1055/s-2008-1073139. PMID 18491247
- [Result] Kroiss M, Quinkler M, Lutz WK, Allolio B, Fassnacht M. Drug interactions with mitotane by induction of CYP3A4 metabolism in the clinical management of adrenocortical carcinoma. Clin Endocrinol (Oxf). 2011 Nov;75(5):585-91. doi: 10.1111/j.1365-2265.2011.04214.x. PMID 21883349
- [Result] Hasegawa E, Nakagawa S, Sato M, Tachikawa E, Yamato S. Effect of polyphenols on production of steroid hormones from human adrenocortical NCI-H295R cells. Biol Pharm Bull. 2013;36(2):228-37. doi: 10.1248/bpb.b12-00627. PMID 23370353
- [Result] Arrighi N, Bodei S, Lucente A, Michel MC, Zani D, Simeone C, Cunico SC, Spano P, Sigala S. Muscarinic receptors stimulate cell proliferation in the human urothelium-derived cell line UROtsa. Pharmacol Res. 2011 Oct;64(4):420-5. doi: 10.1016/j.phrs.2011.06.009. Epub 2011 Jun 28. PMID 21718784
- [Result] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Result] Berruti A, Terzolo M, Sperone P, Pia A, Della Casa S, Gross DJ, Carnaghi C, Casali P, Porpiglia F, Mantero F, Reimondo G, Angeli A, Dogliotti L. Etoposide, doxorubicin and cisplatin plus mitotane in the treatment of advanced adrenocortical carcinoma: a large prospective phase II trial. Endocr Relat Cancer. 2005 Sep;12(3):657-66. doi: 10.1677/erc.1.01025. PMID 16172198
- [Derived] Lagana M, Grisanti S, Ambrosini R, Cosentini D, Abate A, Zamparini M, Ferrari VD, Gianoncelli A, Turla A, Canu L, Terzolo M, Tiberio GAM, Sigala S, Berruti A. Phase II study of cabazitaxel as second-third line treatment in patients with metastatic adrenocortical carcinoma. ESMO Open. 2022 Apr;7(2):100422. doi: 10.1016/j.esmoop.2022.100422. Epub 2022 Mar 7. PMID 35272132